CLINICAL TRIAL: NCT02409576
Title: Pilot Study of Expanded , Activated Haploidentical Natural Killer Cell Infusions for Sarcomas
Acronym: NKEXPSARC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB 2014/00452; CTC1400413 (NUH) (Other: Health Sciences Authority; Singapore); CTC1400412 (KKWCH) (Other: Health Sciences Authority ; Singapore)
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Ewing Sarcoma; Rhabdomyosarcoma
Keywords: EWS; RMS
MeSH Terms: conditions — Sarcoma, Ewing; Rhabdomyosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Expanded, activated NK Cells(NKEXPSARC) (Experimental): Intravenous infusion of expanded, activated NK Cells Donor cell will be expanded and activated in the cGMP compliant TECT lab for 10 to 12 days prior to infusion into the patient.
  Interventions: Biological: Expanded , Activated NK cells

INTERVENTIONS:
Biological: Expanded , Activated NK cells — 1. Chemotherapy - Each patient will receive immunosuppressive chemotherapy before infusion of NK cells.
     Day -7 Cyclophosphamide at 60mg/kg Day -6 Fludarabine at 25mg/m2 daily for 5 days
  2. Radiation - Each patient will receive radiation within 48 hr of NK cell infusion to make the tumor cells more sensitive to NK cell killing Radiation 2Gy
  3. Cytokine support - Each pateint will receive IL-2 to support NK cell activation and expansion in vivo Day -1 alternate day for a total of 6 doses
  4. NK cells - Expanded activated haploidentical NK cells will be infused on day 0.

SUMMARY:
Progress in the treatment of children with leukemia and lymphoma results in high cure rates but progress in the treatment of children and adolescents with solid tumors has been slow. Despite aggressive therapy with multimodality treatment involving surgery, radiation and chemotherapy, about two thirds of the patients with metastatic Ewing sarcoma (EWS), and intermediate and high risk rhabdomyosarcoma (RMS) will relapse. The available second line therapies for relapse are limited and often not effective. There is a dire need to look for treatment options beyond conventional means for the treatment of these patients.

Infusions of allogeneic natural killer (NK) cells in leukemia patients have shown to be tolerated well without inducing graft versus host disease (GVHD). There is also mounting evidence that NK cells have activity against solid tumors.

In the lab the investigators tested NK cell activity against cell lines from different paediatric solid tumors. Among paediatric solid tumors, EWS and RMS are exquisitely sensitive to killing by expanded NK cells; NK cells also have activity against OS cells. Preliminary clinical data suggest that donor NK cells may exert antitumor activity in children with solid tumors undergoing allogeneic hematopoietic stem cell transplantation.

Taking into account the safety of adaptive NK cell infusion, and their efficacy against EWS, RMS and OS, NK cells could be a powerful new tool in the treatment of paediatric solid tumors.

The great anti-tumor activity of expanded and activated NK cells, together with the feasibility of infusing haploidentical NK cells in a non-transplant setting form a compelling rationale for the clinical testing of these NK cells in patients with sarcoma.

DETAILED DESCRIPTION:
Adoptive transfer of allogeneic NK cells has been shown to be safe in patients with leukemia.

The patients enrolled on this will receive lymphodepleting chemotherapy with cyclophosphamide (1 day) followed by fludarabine (5 days) Each patient will receive IL-2 on alternate days starting 1 day before infusion of NK cells for a total of 6 doses.

Patient will undergo imaging MRI or PET or CT scan one month after the infusion to assess response to the NK cell infusion.

In our study we aim to determine the feasibility, safety and efficacy of expanded, activated NK cells in patients with EWS and RMS .

We will also study the persistence and phenotype of expanded NK cells in research participants with EWS and RMS .

The main hypothesis to be tested in this study is that infusion of expanded, activated haploidentical NK cells can produce measurable clinical responses in patients with EWS and RMS .

ELIGIBILITY:
Inclusion Criteria:

A ) NK cell Recipient:

1. Age 0 months to 80 years old.
2. Patients with metastatic, progressive or relapsed EWS, RMS after completing standard of care therapy who are at high risk of relapse even if they do not have any evidence of residual disease.

   a) For patients without residual disease at the point of study entry, response to NK cells will be measured by their incidence of relapse as indicated by their 5-year event free survival. Only patients at high risk of relapse > 70% will be enrolled if there is no evidence of residual disease.
3. Shortening fraction greater than or equal to 25%. Left ventricular ejection fraction (LVEF) greater than or equal to 40%
4. Glomerular filtration rate greater than or equal to 60 ml/min/1.73 m2.
5. Pulse oximetry greater than or equal to 92% on room air.
6. Direct bilirubin less than or equal to 3.0 mg/dL (50 mmol/L).
7. Alanine aminotransferase (ALT) is no more than 2 times the upper limit of normal.
8. Aspartate transaminases (AST) is no more than 2 times the upper limit of normal.
9. Karnofsky or Lansky performance score of greater than or equal to 50.
10. Does not have a current pleural or pericardial effusion.
11. Has a suitable adult family member donor available for NK cell donation.
12. Has recovered from all acute NCI Common Terminology Criteria for Adverse Events (CTCAE) grade II-IV non-hematologic acute toxicities resulting from prior therapy per the judgment of the PI.
13. At least two weeks since receipt of any biological therapy, systemic chemotherapy, and/or radiation therapy.
14. Is not receiving more than the equivalent of prednisone 10 mg daily.
15. Not pregnant (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment).
16. Not lactating.

B) NK cell Donor:

1. First and second degree relative acceptable.
2. 18 years of age or above.
3. Not lactating.
4. Greater than or equal to 3 of 6 HLA match to recipient.
5. Meets eligibility and suitability criteria for hematopoietic cells donation as per institutional guidelines.
6. Not pregnant (negative serum or urine pregnancy test to be conducted within 7 days prior to enrollment).
7. HIV negative. Negative results must be within 60 days prior to enrolment.

Exclusion Criteria:

Failure to meet any of the inclusion criteria.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Disease response after expanded activated NK cell infusion | 1 month post-NK cell infusion (and at regular intervals thereafter till a year post-NK cell infusion)
  Radiological response will be measured based on PET or MRI or CT scan whichever is appropriate imaging for the tumor type and location.

SECONDARY OUTCOMES:
Persistence and phenotype of expanded NK cells in research participants with EWS, RMS and OS. | 1 month ( 30 days) post- NK cell infusion
  NK cell persistence and phenotype will be monitored weekly upto 4 weeks post infusion from peripheral blood.
Toxicity of NK cells infusion (NCI toxicity criteria CTC version 4.0) | 1 month ( 30 days) post- NK cell infusion
  Patients will be monitored for toxicity based on NCI toxicity criteria CTC version 4.0
Performance status will be assessed by age-dependent Performances Scores ( Lansky scale or Karnofsky performance scale) | Initiation of conditioning till 30 days post-NK cell infusion
  Patients performance status will be monitored using Lansky scale for patients below 16 years of age and Karnofsky performance scale for patients more than 16 years of age.
Acute and Chronic GVHD | Initiation of conditioning until 1 month ( 30 days) post- last dose of IL-2
  Patients will monitored for clinical evidence of GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Bernice Oh, Principal Investigator — Department of Paediatrics, National University Hospital; Dario Campana, Principal Investigator — Department of Paediatrics, National University of Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Cho D, Shook DR, Shimasaki N, Chang YH, Fujisaki H, Campana D. Cytotoxicity of activated natural killer cells against pediatric solid tumors. Clin Cancer Res. 2010 Aug 1;16(15):3901-9. doi: 10.1158/1078-0432.CCR-10-0735. Epub 2010 Jun 11. PMID 20542985
- [Background] Perez-Martinez A, de Prada Vicente I, Fernandez L, Gonzalez-Vicent M, Valentin J, Martin R, Maxwell H, Sevilla J, Vicario JL, Diaz MA. Natural killer cells can exert a graft-vs-tumor effect in haploidentical stem cell transplantation for pediatric solid tumors. Exp Hematol. 2012 Nov;40(11):882-891.e1. doi: 10.1016/j.exphem.2012.07.004. Epub 2012 Jul 4. PMID 22771496